CLINICAL TRIAL: NCT07015814
Title: Comparative Evaluation of Glycemic Index of Different Types of Jaggery Produced Locally in Pakistan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rehman Medical Institute - RMI (Other)
Responsible Party: Principal Investigator, Naseer Ahmed, Associate Professor, Rehman Medical Institute - RMI
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GL/GI-NA_1V2
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Glycemic Index and Glycemic Load
Keywords: glycemic index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (cross over) (Active Comparator): Participants will receive all test interventions (2 different varieties of jaggery and a glucose reference) in a randomized sequence with appropriate washout periods between each session. Blood glucose levels will be measured after each test food to determine and compare glycemic index values.
  Interventions: Other: Golden sugarcane jaggery; Other: Dark brown sugarcane jaggery

INTERVENTIONS:
Other: Golden sugarcane jaggery — Participants will consume a standardized portion of jaggery Type A providing 50 grams of available carbohydrates. Capillary blood glucose will be measured over a 2-hour postprandial period.
Other: Dark brown sugarcane jaggery — Participants will consume a standardized portion of jaggery Type B providing 50 grams of available carbohydrates. Capillary blood glucose will be measured over a 2-hour postprandial period.

SUMMARY:
This study aims to evaluate and compare the glycemic index (GI) of various types of jaggery by measuring their effect on blood glucose levels in healthy individuals. Using glucose as the reference standard , the objective is to determine how different jaggery types influence postprandial blood sugar response.

DETAILED DESCRIPTION:
This study aims to evaluate and compare the glycemic index (GI) of various types of jaggery by measuring their effect on blood glucose levels in healthy individuals. Using glucose as the reference standard , the objective is to determine how different jaggery types influence postprandial blood sugar response. The findings will help identify which types of jaggery have lower glycemic impact, contributing to better dietary choices for glycemic control.

ELIGIBILITY:
Inclusion Criteria:Participants should be clinically healthy, as determined by their medical records and verbal history. Only individuals with normal fasting blood glucose levels (70-99 mg/dL) during screening will be eligible -

Exclusion Criteria:1) Participants must not have any chronic disease, not be taking any medications that influence carbohydrate metabolism (such as corticosteroids or metformin), and should be non-smokers and non-alcoholics.

2) Pregnant or lactating female participants, as well as any person with gastrointestinal, metabolic, or endocrine disease (e.g., thyroid disease, PCOS, IBD), will be excluded.

3) Also, subjects with a history of recent acute illness (within the last 2 weeks) will be deferred.

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Glycemic Index (GI) of Different Types of Jaggery | Measured at multiple time points post-consumption (e.g., 0, 15, 30, 45, 60, 90, and 120 minutes) during each test session.
  The incremental area under the blood glucose response curve (iAUC) over 2 hours after consumption of each type of jaggery, expressed as a percentage of the glucose reference.

SECONDARY OUTCOMES:
Postprandial Blood Glucose Response Curve | Same as primary outcome (0-120 minutes).
  Blood glucose levels at each time point following consumption of jaggery types and glucose, to assess the shape and peak of glycemic response.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehman Medical Institue, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fats and oils in human nutrition. Report of a joint expert consultation. Food and Agriculture Organization of the United Nations and the World Health Organization. FAO Food Nutr Pap. 1994;57:i-xix, 1-147. No abstract available. PMID 7641870
- [Background] International Diabetes Federation. (2021). *IDF Diabetes Atlas* (10th ed.). Brussels, Belgium: IDF.
- [Background] Jenkins DJ, Wolever TM, Taylor RH, Barker H, Fielden H, Baldwin JM, Bowling AC, Newman HC, Jenkins AL, Goff DV. Glycemic index of foods: a physiological basis for carbohydrate exchange. Am J Clin Nutr. 1981 Mar;34(3):362-6. doi: 10.1093/ajcn/34.3.362. PMID 6259925